CLINICAL TRIAL: NCT01274390
Title: Impact of Blood Storage Duration on Physiologic Measures: RECESS Ancillary Physiologic Study (RECAP)
Brief Title: Impact of Blood Storage Duration on Physiologic Measures
Acronym: RECAP
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00021198; R01HL101382 (NIH)
Record Dates: First submitted 2011-01-09; First posted 2011-01-11 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2014-07

CONDITIONS: Cardiac Surgery; Erythrocyte Transfusion
Keywords: Cardiac Surgery; Red Blood Cell; Transfusion; Oxygen Saturation; Microvascular Flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Shorter-storage red blood cell units: Red blood cell units stored <= 10 days
- Longer-storage red blood cell units: Red blood cell units stored >= 21 days

SUMMARY:
This study is an ancillary (add-on) study to the clinical trial entitled Red Cell Storage Duration Study (RECESS), which has clinicaltrials.gov identifier NCT00991341. The RECESS study randomizes cardiac surgery patients to receive either red blood cell units stored for no more than 10 days, or red blood cell units stored for at least 21 days, if they need any red blood cell transfusions during their hospital stay for the surgery.

This ancillary study is entitled Impact of Blood Storage Duration on Physiologic Measures: RECESS Ancillary Physiologic Study (RECAP). The hypothesis of the RECAP study is that there will be differences between the two randomized treatment groups in how much the following measurements change, from shortly before a red blood cell transfusion to shortly after a red blood cell transfusion, and from before surgery to 24 hours after surgery:

* Oxygen saturation in the hand
* Oxygen saturation in the brain
* Blood flow in the small blood vessels under the tongue.

The RECAP study will also investigate whether changes in the measurements listed above are associated with clinical outcomes, including

* The Multi-Organ Dysfunction Score
* Death from any cause
* Major cardiac events
* Major pulmonary events

ELIGIBILITY:
Inclusion Criteria:

* Eligible and randomized in the RECESS study (NCT00991341)
* At least 18 years old
* Willing to comply with protocol and provide written informed consent for both RECESS and RECAP
* Scheduled to undergo coronary artery bypass (CABG), valve, or combined CABG plus valve surgery

Exclusion Criteria:

* Prior randomization into the RECESS or RECAP studies
* Undergoing off-pump cardiac surgery
* Undergoing a significant concomitant surgical procedure
* Known sickle cell disease
* Participation in a clinical trial (except observational studies or RECESS) within the previous 30 days
* Received any investigational product within prior 30 days
* Not able to be randomized in RECESS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients enrolled in the RECESS study (NCT00991341) at selected hospitals
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in thenar oxygenation saturation | From a measurement taken within 2 hours prior to the index transfusion, to a measurement taken within 2 hours following the index transfusion.

SECONDARY OUTCOMES:
Change in downslope of thenar oxygen saturation | From a measurement taken within 2 hours prior to the index transfusion, to a measurement taken within 2 hours following the index transfusion.
Change in upslope of thenar oxygen saturation | From a measurement taken within 2 hours prior to the index transfusion, to a measurement taken within 2 hours following the index transfusion.
Change in cerebral oxygenation | From a measurement taken within 2 hours prior to the index transfusion, to a measurement taken within 2 hours following the index transfusion.
Change in microvascular mean flow index | From a measurement taken within 2 hours prior to the index transfusion, to a measurement taken within 2 hours following the index transfusion.
Change in percent perfused vessels | From a measurement taken within 2 hours prior to the index transfusion, to a measurement taken within 2 hours following the index transfusion.
Change in capillary density index | From a measurement taken within 2 hours prior to the index transfusion, to a measurement taken within 2 hours following the index transfusion.
Change in thenar oxygen saturation | From a measurement taken within 6 hours prior to surgery, to a measurement taken 20-28 hours after surgery
Change in downslope of thenar oxygen saturation | From a measurement taken within 6 hours prior to surgery, to a measurement taken 20-28 hours after surgery
Change in upslope of thenar oxygen saturation | From a measurement taken within 6 hours prior to surgery, to a measurement taken 20-28 hours after surgery
Change in cerebral oxygenation | From a measurement taken within 6 hours prior to surgery, to a measurement taken 20-28 hours after surgery
Change in microvascular mean flow index | From a measurement taken within 6 hours prior to surgery, to a measurement taken 20-28 hours after surgery
Change in percent perfused vessels | From a measurement taken within 6 hours prior to surgery, to a measurement taken 20-28 hours after surgery
Change in capillary density index | From a measurement taken within 6 hours prior to surgery, to a measurement taken 20-28 hours after surgery
Change in multi-organ dysfunction score | From pre-surgery baseline to post-operative Day 7, hospital discharge, or death, whichever occurs first
All-cause mortality | Through post-operative Day 28
Composite of major cardiac events | Through post-operative Day 7, hospital discharge, or death, whichever occurs first
Composite of major pulmonary events | Through post-operative Day 7, hospital discharge, or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Bennett-Guerrero, MD, Principal Investigator — Duke University; Christopher Stowell, MD, PHD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Result] Stowell CP, Whitman G, Granger S, Gomez H, Assmann SF, Massey MJ, Shapiro NI, Steiner ME, Bennett-Guerrero E. The impact of red blood cell storage duration on tissue oxygenation in cardiac surgery. J Thorac Cardiovasc Surg. 2017 Mar;153(3):610-619.e2. doi: 10.1016/j.jtcvs.2016.11.029. Epub 2016 Nov 19. PMID 28027790